CLINICAL TRIAL: NCT06655259
Title: An Open-Label, Prospective, Single-Arm Clinical, Phase II Study on the Efficacy and Safety of TURP Combined with Standard Systemic Therapy in Patients with Metastatic Prostate Cancer
Brief Title: Combination of TURP and Standard Systemic Therapy for MPCa
Acronym: CTUSMEP01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ding-Wei Ye, MD, Professor of Urology, Fudan University Cancer Hospital, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2409304-4
Record Dates: First submitted 2024-10-13; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Prostate Cancer
Keywords: mPCa; TURP; ADT; rPFS; prognosis
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Intervention Model Description: This is a single-arm, open-label, prospective Phase II clinical trial. The model focuses on evaluating the combination of TURP (Transurethral Resection of the Prostate) and standard systemic therapy in patients newly diagnosed with metastatic prostate cancer (mPCa). All participants will receive TURP followed by androgen deprivation therapy (ADT), and second-generation anti-androgens such as abiraterone or enzalutamide. The study aims to assess both the efficacy and safety of this combined approach, with radiographic progression-free survival (rPFS) as the primary outcome, and secondary outcomes including overall survival (OS), biochemical progression-free survival (bPFS), and PSA response. The trial is conducted at a single center with a targeted enrollment of 200 patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TURP Combined with Standard Systemic Therapy (Experimental): Participants in this arm will undergo Transurethral Resection of the Prostate (TURP) to alleviate urinary obstruction and reduce tumor burden, followed by Standard Systemic Therapy. This includes Androgen Deprivation Therapy (ADT) with either an LHRH agonist or antagonist, combined with a second-generation anti-androgen, such as abiraterone or enzalutamide, depending on the patient's condition. The goal is to assess the efficacy and safety of this combined approach in treating patients with metastatic prostate cancer (mPCa).
  Interventions: Procedure: TURP; Drug: Standard Medical Therapy

INTERVENTIONS:
Procedure: TURP — Participants will undergo Transurethral Resection of the Prostate (TURP), a surgical procedure performed to relieve symptoms of urinary obstruction caused by the prostate tumor
Drug: Standard Medical Therapy — Participants will receive Standard Medical Therapy, which includes ADT, typically with an LHRH agonist or antagonist, to reduce testosterone levels, a key driver of prostate cancer progression. In addition to ADT, participants may be treated with second-generation anti-androgen drugs such as Abiraterone or Enzalutamide. These medications block androgen receptor signaling and further inhibit the cancer's ability to grow.

SUMMARY:
This is a Phase II, open-label, prospective, single-arm clinical study designed to evaluate the efficacy and safety of combining transurethral resection of the prostate (TURP) with standard systemic therapy in patients with metastatic prostate cancer (mPCa). All participants will undergo TURP to relieve urinary obstruction and reduce tumor burden, followed by androgen deprivation therapy (ADT) and second-generation anti-androgen agents, such as abiraterone or enzalutamide. The primary outcome is radiographic progression-free survival (rPFS), with secondary outcomes including overall survival (OS), biochemical progression-free survival (bPFS), PSA response rates at 3 and 6 months, and quality of life assessments. The trial will enroll 200 newly diagnosed metastatic prostate cancer patients, with regular follow-up for monitoring disease progression and treatment safety. The study will be conducted at Fudan University Cancer Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must voluntarily agree to participate and provide signed informed consent.
2. aged 18 to 80 years.
3. Pathologically or cytologically confirmed adenocarcinoma of the prostate, with neuroendocrine differentiation components ≤10%, and no small cell or signet ring cell carcinoma histological features.
4. Newly diagnosed metastatic prostate cancer with evidence of metastasis (lymph node, bone, or visceral metastases) confirmed by PSMA/PET-CT, CT, or MRI.
5. Patients must not have participated in or plan to participate in another clinical trial.
6. ECOG PS score of 0-1.
7. Adequate Organ and Bone Marrow Function:

   * Absolute neutrophil count (ANC) ≥ 1.5×10⁹/L (1500/μL).

     * Hemoglobin ≥ 90 g/L (9.0 g/dL).

       * Platelet count ≥ 80×10⁹/L (100,000/μL).

         * Liver function: total bilirubin ≤ 1.5×ULN, AST/ALT and alkaline phosphatase ≤ 2.5×ULN.

           Ⅴ. Kidney function: serum creatinine ≤ 2×ULN or calculated creatinine clearance ≥ 30 mL/min.

           Ⅵ. Coagulation function: INR ≤ 1.5.

Exclusion Criteria:

1. History of hypersensitivity or intolerance to any of the drugs used in the study.
2. Patients diagnosed with metastatic castration-resistant prostate cancer (mCRPC) who have already undergone TURP and do not present with lower urinary tract obstruction or hematuria.
3. Oligometastatic mHSPC Patients: Patients with oligometastatic hormone-sensitive prostate cancer (mHSPC) who are planning to undergo radical prostatectomy as the primary treatment.
4. Patients with significant contraindications to TURP, such as severe urethral stricture or inability to catheterize.
5. History of seizures or medications known to lower the seizure threshold, or any disease that may induce seizures (e.g., stroke or transient ischemic attacks) within 12 months prior to the study.
6. Recent Major Surgery: Patients who have undergone major surgery within 4 weeks before starting the study treatment.
7. History of severe or unstable cardiovascular disease within the last 6 months, including severe angina, myocardial infarction, congestive heart failure (NYHA III or higher), cerebrovascular accident, or requiring medication for arrhythmia.
8. Severe Digestive Disorders: Patients with chronic diarrhea, bowel obstruction, or other factors affecting drug absorption.
9. Patients with active infections, including HIV, hepatitis B (HBsAg-positive), or hepatitis C, that may affect the safety and efficacy of the treatment.
10. Patients diagnosed with other malignancies in the past 3 years, excluding cured basal cell carcinoma of the skin.
11. Patients with active brain metastases or leptomeningeal disease.
12. Patients currently receiving any investigational drugs or devices.
13. Patients who are unlikely to comply with the treatment protocol and follow-up schedule.
14. Any condition that the investigator believes could compromise the patient's safety or interfere with the study results (e.g., uncontrolled hypertension, severe diabetes, psychiatric conditions).

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2024-09-21 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Radiographic Progression-Free Survival (rPFS) | 2 years
  Defined as the time from the start of treatment to radiographic evidence of disease progression, assessed by imaging techniques such as PSMA PET-CT, MRI, or CT scans, following RECIST 1.1 criteria. The primary objective is to evaluate how long patients remain free from disease progression after receiving the combination of TURP and standard systemic therapy.
Urinary Symptom Relief Rate | 2 years
  Urinary symptom relief will be assessed using the International Prostate Symptom Score (IPSS) and objective measures like urine flow rate. The goal is to evaluate the extent to which TURP alleviates urinary obstruction and related symptoms in patients with metastatic prostate cancer.

SECONDARY OUTCOMES:
Overall Survival (OS) | 2 years
  Defined as the time from the start of treatment until death from any cause. For patients who are still alive, the time will be censored at the last follow-up. This secondary outcome measure aims to assess the overall survival rate of patients receiving the combination of TURP and standard systemic therapy for metastatic prostate cancer, comparing survival outcomes over the course of the study.
Biochemical Progression-Free Survival (bPFS) | 2 years
  Defined as the time from the start of treatment to biochemical progression, according to the criteria set by the American Society for Radiation Oncology (ASTRO) and the American Urological Association (AUA). Biochemical progression is typically defined as an increase in PSA (Prostate-Specific Antigen) level by 2 ng/mL or more above the nadir (lowest point). This measure will assess how long patients maintain PSA control after receiving the combination of TURP and standard systemic therapy.
3-, 6-Months PSA Response Rate | 3 and 6 months
  The proportion of patients whose Prostate-Specific Antigen (PSA) levels decrease by more than 50% from baseline will be measured at 3 months and 6 months post-treatment. The PSA response rate will be assessed at both time points to evaluate the effectiveness of the combined TURP and standard systemic therapy in reducing PSA levels, which is a key marker of prostate cancer activity.
Quality of Life Assessment | Baseline, 3, 6, 12, and 24 months
  This outcome will evaluate changes in patients' quality of life using the EORTC QLQ-C30 questionnaire. It assesses physical, emotional, and social well-being during and after treatment. The score ranges from 0 to 100, with higher scores indicating a better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China